CLINICAL TRIAL: NCT03208374
Title: Exercise Exposure Data Collection in Patients Undergoing Tumor Molecular Profiling
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17-327
Record Dates: First submitted 2017-07-03; First posted 2017-07-05 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Cancer; Carcinoma
Keywords: Histologically confirmed cancer; IMPACT testing; 17-327
MeSH Terms: conditions — Neoplasms; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MSK-IMPACT genetic panel testing: Participants have completed MSK-IMPACT genetic panel testing on Memorial Sloan Kettering Cancer Center protocol IRB #12-245 and/or IRB #06-107 and/or IRB # 09-141 in the last 3 years.
  Interventions: Behavioral: Prior Exercise Behavior Questions - Harvard Health Professionals Exercise Questionnaire; Behavioral: Current Exercise Behavior Questions: International Physical Activity Questionnaire Short Form (IPAQ SF)

INTERVENTIONS:
Behavioral: Prior Exercise Behavior Questions - Harvard Health Professionals Exercise Questionnaire — Participants will be asked how often on average over the year prior to their most recent diagnosis they participated in walking or hiking; jogging; running; calisthenics, aerobics, rowing, Nordic track; bicycling; tennis, squash, racquetball; lap swimming; weightlifting; and other aerobic exercise (e.g. heavy outdoor work), as well as their usual walking pace and flights of stairs climbed daily over the past 12 months prior to diagnosis.
Behavioral: Current Exercise Behavior Questions: International Physical Activity Questionnaire Short Form (IPAQ SF) — The purpose of this questionnaire is to provide common instruments that can be used to obtain internationally comparable data on exercise exposure in adults aged 15 to 80 years old.
  Other Names: IPAQ SF

SUMMARY:
This study will recruit approximately 5,000 patients with histologically confirmed cancer who have successfully completed MSK-IMPACT panel testing and collect information about tumor genetic results and patient exercise behavior history.

The purpose of the study is to create a registry to collect exercise behavior history in patients who had IMPACT genetic panel testing on protocol IRB #12-245 "Genomic Profiling in Cancer Patients", IRB #06-107 "Storage and Research Use of Human Biospecimens," or IRB #09-141 "Collection of Human Biological Specimens from Patients for Research Studies." The investigators want to find a way to create an exercise database. This database will collect information about tumor genetic results and patient exercise behavior history.

ELIGIBILITY:
Cohort 1: IMPACT Cohort

Inclusion Criteria:

* Histologically-confirmed cancer.
* IMPACT testing with completed genomic profile completed within three years of initial recruitment approach
* Registered to Memorial Sloan Kettering Cancer Center protocol IRB# 12-245 and/or IRB #06-107 and/or IRB # 09-141
* ≥ 18 years of age
* ECOG Performance Status of 0 or 1

Exclusion Criteria:

* Unable to speak and read English
* Not willing to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study cohort will consist of approximately 5,000 participants with histology confirmed cancer who have successfully completed MSK-IMPACT panel testing and are being treated at any Memorial Sloan Kettering Cancer Center site.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Characterize exercise participant behavior history via exercise survey | Up to 5 years
  Participants who have undergone MSK-IMPACT panel testing will complete the exercise history survey. The 10 minute survey only asks participants about their exercise history, both in period before their most recent diagnosis as well as their current exercise behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org